CLINICAL TRIAL: NCT02774525
Title: Concurrent Treatment of Substance Abuse and Child Maltreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Ron Prinz, PhD, Carolina Distinguished Professor, University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00015175
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Substance Use; Child Maltreatment
Keywords: child welfare system; parental substance use problem; child maltreatment; parenting
MeSH Terms: conditions — Substance-Related Disorders | interventions — Pharmaceutical Preparations; Ethanol; Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment as Usual (TAU) (Active Comparator): Outpatient substance-abuse treatment plus drug and alcohol screening plus brief support for personal goal setting
  Interventions: Behavioral: Treatment as usual (TAU)
- Contingency Management (Experimental): Contingency management for drug and alcohol abstinence plus TAU
  Interventions: Behavioral: Reinforcement for drug & alcohol abstinence; Behavioral: Treatment as usual (TAU)
- Parenting Intervention (Experimental): Parenting intervention plus TAU
  Interventions: Behavioral: Parenting intervention; Behavioral: Treatment as usual (TAU)
- Parenting Intervention + Contingency Management (Experimental): Parenting intervention plus contingency management for drug and alcohol abstinence plus TAU
  Interventions: Behavioral: Reinforcement for drug & alcohol abstinence; Behavioral: Parenting intervention; Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Reinforcement for drug & alcohol abstinence
  Other Names: Contingency management for negative drug & alcohol samples
  Arms: Contingency Management; Parenting Intervention + Contingency Management
Behavioral: Parenting intervention
  Other Names: Pathways Triple P
  Arms: Parenting Intervention; Parenting Intervention + Contingency Management
Behavioral: Treatment as usual (TAU) — Outpatient substance-abuse therapy plus drug & alcohol screening plus support for personal goal setting

SUMMARY:
The co-occurrence of child maltreatment and parental substance-use problems is a major public health problem with serious consequences for children, parents, families, and the community at large. The need for effective dual treatment of caregiver substance abuse and child maltreatment is unquestionable, but there is a dearth of controlled treatment outcome studies with substance-using parents who have engaged in child maltreatment. This project examines two evidence-based treatments-Contingency Management for substance-use problems and Pathways Triple P parenting intervention to improve parenting for prevention of child-maltreatment recurrence. These two systematic interventions are being tested in the context of traditional outpatient treatment for substance-use problems.

ELIGIBILITY:
Inclusion Criteria:

* open child protective services case for child maltreatment
* beginning intensive outpatient treatment for drug or alcohol use problem
* at least one child 2-8 years of age

Exclusion Criteria:

* not primary custodial parent for child 2-8 years of age
* serious mental illness
* residing outside the two participating counties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
longest duration of negative urine and breath samples | 13 weeks
recurrence of child maltreatment--child protective services records | 18 months after baseline

SECONDARY OUTCOMES:
self-reported substance use--Addiction Severity Index-Lite | 4 months after baseline; 12 months after baseline; 18 months after baseline
  Drug and Alcohol Composite (severity)
parent report of child behavior problems--child behavior inventory | 4 months after baseline; 12 months after baseline; 18 months after baseline
  Intensity score for child behavior problems
self-reported parenting--Parenting Scale; Parenting Practices Interview | 4 months after baseline; 12 months after baseline; 18 months after baseline
  Parenting Scale: Overreactivity; Laxness Parenting Practices Interview: Appropriate Discipline; Harsh and Inconsistent Discipline

OTHER OUTCOMES:
self-reported quality of life--Quality of Life Inventory | 4 months after baseline; 12 months after baseline; 18 months after baseline
self-reported HIV behavioral risk--HIV Risk Behavior Scale | 4 months after baseline; 12 months after baseline; 18 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ron Prinz, Ph.D., Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina Parenting & Family Res Center, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No